CLINICAL TRIAL: NCT04849988
Title: A Phase 2, Randomized, Double-Blind, Multicenter, Placebo Controlled Study to Evaluate the Safety and Efficacy of Intramuscular ABP-450 (prabotulinumtoxinA) Injection for the Treatment of Cervical Dystonia
Brief Title: A Phase 2 Study to Evaluate the Safety and Efficacy of ABP-450 in the Treatment of Cervical Dystonia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AEON Biopharma, Inc. (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ABP-19000
Record Dates: First submitted 2021-04-14; First posted 2021-04-20 (Actual); Results first posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-01

CONDITIONS: Cervical Dystonia
MeSH Terms: conditions — Torticollis | interventions — prabotulinumtoxin A; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Approximately 60 patients will be randomized in a 1:1:1:1 ratio and receive one of the four treatments: ABP-450 low dose, ABP-450 mid dose, ABP-450 high dose, or placebo via intramuscular injection into affected neck muscles.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The investigator, study nurse/other study personnel, and patients will be blinded to the treatment group. An appropriately trained person will reconstitute investigational product, fill masked syringes and provide them to the blinded investigator, but will not perform any assessments with the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ABP-450 - Low Dose (Experimental): ABP-450 Low Dose - Intramuscular injections into affected neck muscles.
  Interventions: Drug: ABP-450
- ABP-450 - Medium Dose (Experimental): ABP-450 Mid Dose - Intramuscular injections into affected neck muscles.
  Interventions: Drug: ABP-450
- ABP-450 - High Dose (Experimental): ABP-450 High Dose - Intramuscular injections into affected neck muscles.
  Interventions: Drug: ABP-450
- Placebo (Placebo Comparator): Placebo (0.9% saline, sterile, unpreserved, USP/Ph.Eur.) - Intramuscular injections into affected neck muscles.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ABP-450 — ABP-450 (prabotulinumtoxinA) contains a 900kDA botulinum toxin type-A complex produced by the bacterium Clostridium botulinum.
  Other Names: prabotulinumtoxinA
  Arms: ABP-450 - High Dose; ABP-450 - Low Dose; ABP-450 - Medium Dose
Drug: Placebo — 0.9% sodium chloride, sterile, unpreserved, USP/Ph.Eur.
  Other Names: 0.9% sodium chloride; saline
  Arms: Placebo

SUMMARY:
This Phase 2 trial will evaluate the safety and efficacy of ABP-450 for the treatment of cervical dystonia in adults. The study will enroll 60 patients across approximately 30 sites in the United States. Study subjects will be divided evenly across a low dose group, a medium dose group, a high dose group, and a placebo group for one treatment cycle.

DETAILED DESCRIPTION:
This Phase 2 trial will evaluate the safety and efficacy of ABP-450 for the treatment of cervical dystonia in adults. The study will enroll 60 patients across approximately 30 sites in the United States. Study subjects will be divided evenly across a low dose, a medium dose group, a high dose and placebo group for one treatment cycle.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients between 18 and 75 years of age (inclusive)
2. A clinical diagnosis of cervical dystonia (ie, spasmodic torticollis) defined by:

   * TWSTRS total score ≥20
   * TWSTRS severity score ≥10
   * TWSTRS disability score ≥3
   * TWSTRS pain score ≥1
3. On a stable dose of medications (if any) used for focal dystonia treatment (eg, anticholinergics and benzodiazepines) for at least 3 months prior to and expected throughout the study duration
4. For pre-treated patients only: Source documentation (eg, patient history) of the last 2 consecutive injection sessions with a botulinum toxin type A
5. For pre-treated patients only: At least 16 weeks must have passed between the last injection with botulinum toxin for cervical dystonia and baseline treatment (patients can be screened at Week 15 but cannot be enrolled until 16 weeks [for Day 0 injection])
6. Provided written informed consent to being treated for cervical dystonia with ABP-450
7. Stated willingness to comply with all study procedures, including attendance at the study center for all study visits as scheduled and have technological capabilities to have televisits

Exclusion Criteria:

1. Traumatic torticollis or tardive torticollis
2. Predominant retrocollis or anterocollis
3. Myotomy or denervation surgery in the affected muscles (eg, peripheral denervation and/or spinal cord stimulation)
4. Hypersensitivity to human serum albumin, sucrose, or botulinum toxin type A
5. Previous treatment for cervical dystonia with rimabotulinumtoxin B
6. Diagnosis of myasthenia gravis, Lambert-Eaton syndrome, amyotrophic lateral sclerosis, or any other significant neuromuscular disease that might interfere with the trial
7. Current swallowing disorder of any origin (dysphagia scale ≥3, ie, severe, with swallowing difficulties and requiring a change in diet)
8. Marked limitation on passive range of motion that suggests contractures or other structural abnormality, eg, cervical contractures or cervical spine syndrome
9. Treatment with botulinum toxins of any type for any indication other than cervical dystonia within 16 weeks prior to baseline and during the study
10. Medical or psychiatric conditions that may increase the risk associated with study participation or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study
11. Participation in another interventional study during participation in this study
12. Pregnant or lactating females, or females of child-bearing potential not willing to use an acceptable method of contraception (ie, intrauterine device, barrier methods with spermicide, or abstinence)
13. For pre-treated patients only: The patient's most recent injection with botulinum toxin exceeding the number of units specified as follows:

    * OnabotulinumtoxinA (BOTOX®): >300 units
    * IncobotulinumtoxinA (Xeomin®): >300 units
    * AbobotulinumtoxinA (Dysport®): >750 units

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2022-07-11 (Actual); Study Completion 2022-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Comella, MD, Principal Investigator — Rush University Medical Center; Joseph Jankovic, Principal Investigator — Baylor St. Luke's Medical Center
Locations (21):
- United States (21):
  - Arizona Neuroscience Research, Phoenix, Arizona
  - Movement Disorder Center of Arizona, Scottsdale, Arizona
  - Parkinson's and Movement Disorder Institute, Fountain Valley, California
  - Neuro Pain Medical Center, Fresno, California
  - Loma Linda University, Loma Linda, California
  - New England Institute for Neurology and Headache, Stamford, Connecticut
  - Infinity Clinical Research LLC, Hollywood, Florida
  - The Neurology Research Group, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Neurology One, Winter Park, Florida
  - Emory University, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Michigan State University, East Lansing, Michigan
  - Quest Research Institute - Hunt - PPDS, Farmington Hills, Michigan
  - University of New Mexico, Albuquerque, New Mexico
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Cleveland Clinic Lou Ruvo Center for Brain Health, Cleveland, Ohio
  - The Orthopedic Foundation, New Albany, Ohio
  - Veracity Neuroscience LLC, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data collected during the trial, after deidentification may be shared following review of the clinical study report by the FDA review division and if a decision is made to publish the results in a publication outside posting the results in clinicaltrials.gov.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 25 sites in the U.S. between March 29, 2021 and July 11, 2021.
Pre-assignment Details: Of the 70 participants screened, 61 were randomized. There were 59 participants randomized and dosed, and 57 of them were included in the modified full analysis set (mFAS) for the efficacy analysis.
Groups:
- Placebo: Placebo (0.9% unpreserved saline) - Intramuscular injections into affected neck muscles.
- ABP-450 - 150U: ABP-450 Low Dose - Intramuscular injections into affected neck muscles.
- ABP-450 - 250U: ABP-450 Medium Dose - Intramuscular injections into affected neck muscles.
- ABP-450 - 350U: ABP-450 High Dose - Intramuscular injections into affected neck muscles.
Period: Overall Study
Arm/Group | Placebo | ABP-450 - 150U | ABP-450 - 250U | ABP-450 - 350U
Started (Two participants were randomized in error, but they were not dosed due to failure to meet eligibility criteria.) | 15 | 15 | 16 | 15
Randomized But Not Dosed | 1 | 1 | 0 | 0
Treated | 14 | 14 | 16 | 15
Safety Analysis Set (For this row and below, the number of participants in the Safety Analysis Set is used as the denominator for percentages.) | 14 | 14 | 16 | 15
Full Analysis Set | 14 | 14 | 16 | 15
Modified Full Analysis Set (Two participants were excluded from the modified Full Analysis Set due to a change in their background medication.) | 14 | 14 | 14 | 15
Completed | 11 | 9 | 13 | 10
Not Completed | 4 | 6 | 3 | 5
Not completed — Lack of Efficacy | 3 | 4 | 1 | 4
Not completed — Other reasons | 1 | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Two patients were excluded from the analysis due to a change in their background medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | ABP-450 - 150U | ABP-450 - 250U | ABP-450 - 350U | Total
Number analyzed (Participants) | 14 | 14 | 14 | 15 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (11.06) | 55.8 (12.97) | 54.6 (13.61) | 55.3 (11.39) | 56.2 (12.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 13 | 12 | 39
  Male | 7 | 7 | 1 | 3 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 0 | 2
  White | 13 | 14 | 11 | 14 | 52
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1 | 2
Previous treatment with BOTOX® [Count of Participants; unit: Participants] | 10 | 9 | 11 | 10 | 40
Duration of Cervical Dystonia [Mean (Standard Deviation); unit: years] | 14.83 (11.134) | 14.58 (10.799) | 7.36 (6.464) | 11.53 (7.175) | 12.26 (9.421)
Baseline TWSTRS-Total Score [Mean (Standard Deviation); unit: units on a scale] | 39.68 (7.525) | 44.30 (6.093) | 42.20 (11.585) | 43.62 (9.847) | 42.47 (8.962)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Related Serious Adverse Events
Description: The primary safety endpoint will be the number of participants with treatment-related serious adverse events since the start of treatment by Treatment Group when dosed with placebo, ABP-450 (low dose), ABP-450 (medium d dose), or ABP-450 (high dose).
Time Frame: Baseline up to 20 Weeks
Population: All treated patients are accounted for in the Treatment-related Serious Adverse Events data table including the two patients with changes in background medications.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ABP-450 - 150U | ABP-450 - 250U | ABP-450 - 350U
Number analyzed (Participants) | 14 | 14 | 16 | 15
Participants | 0 | 0 | 0 | 0

2. Secondary Outcome: Mean Change of the Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS)-Total Score From Baseline to Week 4
Description: The Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) scale is used to assess the severity of cervical Dystonia. The TWSTRS-total score has a minimum score of 0 and a maximum score of 85, where higher scores represent worse outcomes. It comprises 3 subscales, which are summated to get the total score: the Torticollis Severity Scale (minimum score of 0, maximum score of 35), the Disability Scale (minimum score of 0, maximum score of 30), and the Pain Scale (minimum score of 0, maximum score of 20).
Time Frame: Baseline to Week 4
Population: Two patients were excluded from the analysis due to a change in their background medication.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ABP-450 - 150U | ABP-450 - 250U | ABP-450 - 350U
Number analyzed (Participants) | 14 | 14 | 14 | 15
score on a scale | 3.57 (2.67) | 14.01 (2.63) | 11.28 (2.70) | 9.92 (2.54)

3. Secondary Outcome: Mean Change in the Subscale Score of Disability of the Baseline Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) From Baseline to Week 4
Description: The Disability subscale of the Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) is used to assess the severity of disability in cervical dystonia. The disability subscale has a minimum score of 0 and maximum score of 30, where higher scores represent worse outcomes.
Time Frame: Baseline to Week 4
Population: Two patients were excluded from the analysis due to a change in their background medication.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ABP-450 - 150U | ABP-450 - 250U | ABP-450 - 350U
Number analyzed (Participants) | 14 | 14 | 14 | 15
score on a scale | 1.02 (1.11) | 4.53 (1.09) | 4.24 (1.14) | 2.62 (1.06)

4. Secondary Outcome: Mean Change in the Subscale Score of Pain of the Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) From Baseline to Week 4
Description: The Pain subscale of the Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) is used to assess the severity of pain in cervical dystonia. The pain subscale has a minimum score of 0 and maximum score of 20, where higher scores represent worse outcomes.
Time Frame: Baseline to Week 4
Population: Two patients were excluded from the analysis due to a change in their background medication.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ABP-450 - 150U | ABP-450 - 250U | ABP-450 - 350U
Number analyzed (Participants) | 14 | 14 | 14 | 15
score on a scale | 1.27 (1.10) | 3.56 (1.05) | 3.58 (1.08) | 3.69 (1.02)

5. Secondary Outcome: Mean Change in the Subscale Score of Severity of the Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) From Baseline to Week 4
Description: The Severity subscale of the Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) is used to assess the severity of torticollis in cervical dystonia. The severity subscale has a minimum score of 0 and maximum score of 35, where higher scores represent worse outcomes.
Time Frame: Baseline to Week 4
Population: Two patients were excluded from the analysis due to a change in their background medication.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | ABP-450 - 150U | ABP-450 - 250U | ABP-450 - 350U
Number analyzed (Participants) | 14 | 14 | 14 | 15
score on a scale | 1.91 (0.91) | 5.89 (0.91) | 2.94 (0.97) | 3.45 (0.87)

6. Secondary Outcome: Mean Change in Patient Global Impression of Change (PGI-C) From Baseline to Week 4
Description: The PGI-C enables the patient to rate changes in their perception of their general health status over the duration of the assessment via a 7-point scale ranging from "much improved" to "much worse". The 7-point scale range is much improved (+3) to much worse (-3) with no change at "0".
  The mean change in the subject's assessment of the change in clinical status since the start of treatment measured by the Patients' Global Impression of Change (PGI-C) Scale was assessed by Treatment Group at Week 4.
Time Frame: Baseline to Week 4
Population: Two patients were excluded from the analysis due to a change in their background medication.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | ABP-450 - 150U | ABP-450 - 250U | ABP-450 - 350U
Number analyzed (Participants) | 14 | 14 | 14 | 15
units on a scale | 4.0 (1.11) | 2.6 (0.31) | 2.2 (0.32) | 2.7 (0.30)

7. Secondary Outcome: Mean Change in Clinical Global Impression of Change (CGI-C) From Baseline to Week 4
Description: The CGI-C enables the patient to rate changes in their perception of their general health status over the duration of the assessment via a 7-point scale ranging from "much improved" to "much worse". The 7-point scale range is much improved (+3) to much worse (-3) with no change at "0".
  The mean change from Baseline in the Clinical Global Impression of Change (CGI-C) Score was assessed by Treatment Group at Week 4.
Time Frame: Baseline to Week 4
Population: Two patients were excluded from the analysis due to a change in their background medication.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | ABP-450 - 150U | ABP-450 - 250U | ABP-450 - 350U
Number analyzed (Participants) | 14 | 14 | 14 | 15
units on a scale | 3.9 (0.33) | 2.3 (0.32) | 2.0 (0.33) | 2.7 (0.31)

ADVERSE EVENTS:
Time Frame: Up to Week 20
Arm/Group | Placebo | ABP-450 - 150U | ABP-450 - 250U | ABP-450 - 350U
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 9/14 | 8/14 | 12/16 | 11/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=14) | ABP-450 - 150U (N=14) | ABP-450 - 250U (N=16) | ABP-450 - 350U (N=15)
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 2 | 3
Muscular Weakness (Gastrointestinal disorders) | 0 | 2 | 1 | 1
Headache (Nervous system disorders) | 1 | 2 | 2 | 1
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 2 | 1
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0
Head discomfort (Nervous system disorders) | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1
Feeling abnormal (General disorders) | 0 | 0 | 1 | 0
Injection site pain (General disorders) | 1 | 1 | 0 | 0
Injection site pruritus (General disorders) | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0
Diplopia (Eye disorders) | 0 | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 1 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Data are the property of the sponsor and cannot be published without prior authorization from the sponsor.

DOCUMENTS (2):
  • Study Protocol (2021-05-13): https://cdn.clinicaltrials.gov/large-docs/88/NCT04849988/Prot_002.pdf
  • Statistical Analysis Plan (2022-07-22): https://cdn.clinicaltrials.gov/large-docs/88/NCT04849988/SAP_003.pdf